CLINICAL TRIAL: NCT02230397
Title: Efficacy and Tolerance Evaluation of a Topical "Revitalizing" Face Day Cream: Comparison Within Subjects Versus Placebo
Brief Title: Efficacy and Tolerance Evaluation of a Topical "Revitalizing" Face Day Cream
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Derming SRL (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: E2713
Record Dates: First submitted 2014-07-10; First posted 2014-09-03 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
Keywords: skin aging; anti-aging cream; wrinkles
MeSH Terms: interventions — plantaricin A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- plantaricin a (active product) (Other): Volunteers applied the active product for an uninterrupted period of 8 weeks (on the right or on the left face side randomly) twice a day, in the morning and in the evening, with a mild massage.
  Interventions: Other: plantaricin a (active product)
- placebo product (Other): Volunteers applied the placebo product for an uninterrupted period of 8 weeks (on the right or on the left face side randomly) twice a day, in the morning and in the evening, with a mild massage
  Interventions: Other: placebo product

INTERVENTIONS:
Other: plantaricin a (active product) — Product application: 8 weeks (one on the right and one on the left face side randomly) twice a day, in the morning and in the evening, with a mild massage
  Arms: plantaricin a (active product)
Other: placebo product — Product application: 8 weeks (one on the right and one on the left face side randomly) twice a day, in the morning and in the evening, with a mild massage
  Arms: placebo product

SUMMARY:
Aim of the study was to evaluate clinically and by non-invasive instrumental evaluations the "revitalizing" activity of a face cream applied twice a day, morning and evening, for an uninterrupted period of 8 weeks, by healthy female volunteers aged 45-55 years with face ritidosis and women aged 55-65 years not habitual user of antiage-creams.

The study foresaw the comparison within subjects of the study product versus placebo (half face method).

It was also aim of this study to evaluate products efficacy and cosmetic acceptability by the volunteers and tolerance both by investigator and volunteers.

ELIGIBILITY:
Inclusion Criteria:

* female healthy subjects
* age 45-55 years
* women aged 55-65 years who are not habitual user of antiage-creams
* presence of moderate face ritidosis
* agreeing to present at each study visit without make-up
* accepting to not change their habits regarding food, physical activity, face cleansing and make- up use
* accepting not to expose their face to strong UV irradiation (UV session, or sun bathes) during the entire duration of the study
* accepting to sign the Informed consent form

Exclusion Criteria:

* pregnancy
* lactation
* change in the normal habits regarding foods, physical activity, face cleansing and make-up use during the month preceding the test
* sensitivity to the test products or theirs ingredients
* subjects whose insufficient adhesion to the study protocol is foreseeable
* participation in a similar study actually or during the previous 3 months
* change in the normal life habits during the month preceding the inclusion
* dermatological disease (dermatitis; presence of cutaneous disease on the tested area, as lesions, scars, malformations; recurrent facial/labial herpes)
* clinical and significant skin condition on the test area (e.g. active eczema, dermatitis, psoriasis etc.)
* diabetes
* endocrine disease
* hepatic disorder
* renal disorder
* cardiac disorder
* pulmonary disease
* cancer
* neurological or psychological disease
* inflammatory/immunosuppressive disease
* drug allergy
* drugs/cutaneous medical or surgical procedures at level of the tested area during the previous 3 months
* anti-inflammatory drugs, anti-histaminic, topic and systemic corticosteroids, narcotic, antidepressant, immunosuppressive drugs (with except of contraceptive or hormonal treatment starting from at least 1 year);
* assumption of drugs able to influence the test results in the investigator opinion

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2013-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Profilometry: change from baseline (T4 and T8 vs. T0) | T0 (basal conditions), T4 and T8 (after 4 and 8 week-treatment)
  A picture of crow's feet area was taken thanks to Primos compact portable device (GFMesstechnik); a software able to elaborate 3D representations of skin wrinkles as well as to measure skin principal profilometric parameters in vivo or on skin replicas, according to the law DIN EN ISO 4228; moreover the software compares directly the different images obtained at the times foresee by the protocol (T0, T4 and T8).The portable probe assures a constant distance from the skin as well as a fixed illumination angle of incidence; in this way is possible to acquire standardized and reproducible images.

SECONDARY OUTCOMES:
Skin electrical capacitance: change from baseline (T4 and T8 vs. T0) | T0 (basal condition), T4 and T8 (after 4 and 8 week-treatment)
  Hydration is measured by the instrument Corneometer CM825 (Courage - Khazaka, Köln, Germany): a square sensor (49mm2) frontally covered by a special glass, mounted on a spring cursor able to measure electrical capacity. Leaning the sensor on the skin surface, with a constant pressure thanks to the spring cursor it is possible to perform measures. The sensor acts as a capacitor. When a voltage is applied to this capacitor, the quantity of electric charge stored will be dependent on the dielectric properties of the material in contact with the probe. Water has an unusually high dielectric constant and so its presence in the skin is readily detectable by this method. So the measure of the skin capacitance properties is an indirect expression of its hydration level. To reduce the variability of measurement methods, for each evaluated side, three measures on the same skin area were executed: the adjusted mean will be considered as the real measure value.
Skin plastoelasticity: change from baseline (T4 and T8 vs. T0) | T0 (basal condition), T4 and T8 (after 4 and 8 week-treatment)
  Skin plastoelasticity is measured with the instrument Dermal Torque Meter (Dia-Stron Ltd., UK). This instrument is based on the principle of the torsion given to the skin surface by a probe made of two circles that adhere to the skin through shaped adhesive tapes. The internal circle rotation, while the external circle is still, exerts a constant torsion of the skin (torsion time = 1 second with a torque = 9mN*m). The instrument measures the torsion angle (θ) during the mechanical stimulus ("torque on") and after it has ceased ("torque off").For each of the considered curves the cutaneous rotational ratio relative to defined measured times can be measured, obtaining the parameters listed below:
  Ue: immediate extensibility ("torque on" at 0.02 sec.) Uf: maximum extensibility ("torque on" at 0.9 sec.) Uv: viscoelasticity Ur: immediate elastic recovery ("torque off" at 0.02 sec.).
Spectophotometry: change from baseline (T4 and T8 vs. T0) | T0 (basal condition), T4 and T8 (after 4 and 8 week-treatment)
  Skin colour was measured by a visible-UV-IR (λ from 300 to 900 nm) spectrophotometer which use a tungsten halogen lamp and a deuterium lamp in accordance with CIE (Commission Internationale de l'Eclarage), the main international organisation concerned with colour and colour measurement. Lamps were switched on 30 minutes before instrument use in order to join a stable emission. Measurement angle was 90° (position of the probe on the skin) and measured area was 2 mm2; used wavelength range was 380-780 nm corresponds to the visible light spectrum.
Optical colorimetry: change from baseline (T4 and T8 vs. T0) | T0 (basal condition), T4 and T8 (after 4 and 8 week-treatment)
  Measurement of skin brightness was performed by a tri-stimulus colorimeter (Chroma Meter CR-200®) equipped with three special filters to obtain R,G,B values in accordance with CIE (Commission Internationale de l'Eclarage), the main international organisation concerned with colour and colour measurement. CIE L*a*b* system (CIELAB) is the most complete colour-space specified by the CIE (1976). It describes all the colours visible to the human eye; the three coordinates of L*a*b* represent the lightness of the colour (L* = 0 yields black and L* = 100 indicates diffuse white; specular white may be higher), its position between red/magenta and green (a*, negative values indicate green while positive values indicate magenta) and its position between yellow and blue (b*, negative values indicate blue and positive values indicate yellow).
Tape stripping: | T0 (basal conditions), T4 and T8 (after 4 and 8 week-treatment)
  Tape stripping was performed at each study time on the forehead on 10 selected subjects. The skin was not cleaned before tape stripping and tested area were marked with a black washable pencil. D-squame® discs (Monaderm, Monaco) with a diameter of 22mm were placed on the site of application (area without hair), applied with a constant pressure for 15 sec and then peeled off. The first two strips were discharged. Third and fourth strip were collected and stored at -20°C until following analysis listed below:
  * protein extraction and quantification
  * microscopic analysis
  * study of the expression of biological markers associated with skin ageing
  * study of ageing/oxidative stress
Clinical evaluations: change from baseline (T4 and T8 vs. T0) | T0 (basal conditions), T4 and T8 (after 4 and 8 week-treatment)
  The following clinical evaluations were performed:
  wrinkles grade (nasolabial folds and "crow's feet"): 0 = no wrinkles; 1= very weak wrinkles; 2 = weak wrinkles; 3= quite evident wrinkles; 4 = evident wrinkles; 5 = very evident wrinkles; 6 = marked wrinkles; 7 = very marked wrinkles submental ptosis, scored from 0 (absence of ptosis - very regular oval face) to 5 (very marked ptosis - very irregular oval face) according to a clinical photographic scale.
  surface microrelief: 1 = very regular; 2 = regular; 3 = irregular; 4 = very irregular skin dullness (overall face): 1= luminous skin;2 = normal skin; 3= opaque skin; 4= very opaque skin skin resistance to pinching, to traction and recovery after pinching (malar region): 0 = very important;1 = important; 2 = moderate; 3 = weak; 4 = very weak skin dryness (malar region): 0 = very hydrated skin; 1= hydrated skin; 2 = normal skin; 3= kindly dry skin; 4= dry skin ; 5= very dry skin
Photographic documentation: | T0 (basal condition), T4 and T8 (after 4 and 8 week-treatment)
  In basal condition (T0), at T4 and at T8 the investigator took lateral pictures of each volunteer. In order to assure comparable images, the pictures were taken with standardised methods, concerning especially:
  magnification factor intensity of illumination source (photographic lamps) angle of incidence and inclination of illumination Thanks to the application "remote trigger" (Canon EOS utility software) it was possible to overlay the first photographic image (T0) with the ones taken in the following times (T4 and T8); so it was possible to have totally comparable images.

CONTACTS AND LOCATIONS:
Overall Officials: Adele Sparavigna, Doctor, Principal Investigator — Derming SRL
Locations (1):
- DermIng SRL, Monza, Monza, Italy

REFERENCES:
- [Background] Ascher B, Coleman S, Alster T, Bauer U, Burgess C, Butterwick K, Donofrio L, Engelhard P, Goldman MP, Katz P, Vleggaar D. Full scope of effect of facial lipoatrophy: a framework of disease understanding. Dermatol Surg. 2006 Aug;32(8):1058-69. doi: 10.1111/j.1524-4725.2006.32230.x. PMID 16918569
- [Background] Bradford MM. A rapid and sensitive method for the quantitation of microgram quantities of protein utilizing the principle of protein-dye binding. Anal Biochem. 1976 May 7;72:248-54. doi: 10.1016/0003-2697(76)90527-3. No abstract available. PMID 942051
- [Background] De Jongh CM, Verberk MM, Withagen CE, Jacobs JJ, Rustemeyer T, Kezic S. Stratum corneum cytokines and skin irritation response to sodium lauryl sulfate. Contact Dermatitis. 2006 Jun;54(6):325-33. doi: 10.1111/j.0105-1873.2006.00848.x. PMID 16787454
- [Background] De Rigal J, Leveque JL In vivo measurement of the stratum corneum elasticity Bioengineering and the skin 1: 13-23, 1985
- [Background] Elsner P, Berardesca E, Maibach H Bioengineering of the skin: Water and the stratum corneum CRC Press, Boca Raton, 1994
- [Background] Elsner P, Barel AO, Berardesca E, Gapard B, Serup J Skin Bioengineering Techniques and Applications in Dermatology and Cosmetology Karger, 1998
- [Background] Fernay, Voltaire The World Medical Association (1989) "World Medical Association Declaration of Helsinki", Hong-Kong.
- [Background] Fullerton A, Fischer T, Lahti A, Wilhelm KP, Takiwaki H, Serup J. Guidelines for measurement of skin colour and erythema. A report from the Standardization Group of the European Society of Contact Dermatitis. Contact Dermatitis. 1996 Jul;35(1):1-10. doi: 10.1111/j.1600-0536.1996.tb02258.x. PMID 8896947
- [Background] Frankowsky G., Hainich R., GFMesstechnik GmbH Germany DLP-Based 3D metrology by structured light or projected fringe technology for life sciences and industrial metrology Proc. SPIE Photonics West: 1-12, 2009
- [Background] Garcia Ortiz P, Hansen SH, Shah VP, Menne T, Benfeldt E. Impact of adult atopic dermatitis on topical drug penetration: assessment by cutaneous microdialysis and tape stripping. Acta Derm Venereol. 2009;89(1):33-8. doi: 10.2340/00015555-0562. PMID 19197539
- [Background] Glogau RG. Aesthetic and anatomic analysis of the aging skin. Semin Cutan Med Surg. 1996 Sep;15(3):134-8. doi: 10.1016/s1085-5629(96)80003-4. PMID 8948530
- [Background] Grove GL, Grove MJ, Leyden JJ. Optical profilometry: an objective method for quantification of facial wrinkles. J Am Acad Dermatol. 1989 Sep;21(3 Pt 2):631-7. doi: 10.1016/s0190-9622(89)70230-9. PMID 2778127
- [Background] Grove GL, Zerweck CR, Houser TP, Smith GE, Koski NI. A randomized and controlled comparison of gentleness of 2 medical adhesive tapes in healthy human subjects. J Wound Ostomy Continence Nurs. 2013 Jan-Feb;40(1):51-9. doi: 10.1097/WON.0b013e318276f2a4. PMID 23202590
- [Background] Hoppe U, Sauermann G, Lunderstadt R Quantitative analysis of the skin surface by means of digital signal processing J Soc Cosmet Chem 36: 105-123, 1985
- [Background] Hof, C., Hopermann, H.: University of the Federal Armed Forces, Hamburg Comparison of Replica - and In Vivo - Measurement of the Microtopography of Human Skin
- [Background] Jaspers S., Bretschneider T., Maerkeer U., Ennen J. Optical topometry with Primos: a powerful tool to prove the efficacy on skin care products in in-vivo studies XXI IFSCC International Congress Proceeding, 430-434
- [Background] Jaspers S., Hopermann H. et all Rapid in vivo measurement of the topography of human skin by active image triangulation using a digital micromirror device Skin Research and Technology 5: 195-207, 2006
- [Background] Lademann J, Meinke MC, Schanzer S, Richter H, Darvin ME, Haag SF, Fluhr JW, Weigmann HJ, Sterry W, Patzelt A. In vivo methods for the analysis of the penetration of topically applied substances in and through the skin barrier. Int J Cosmet Sci. 2012 Dec;34(6):551-9. doi: 10.1111/j.1468-2494.2012.00750.x. Epub 2012 Sep 25. PMID 22957937
- [Background] Lademann J, Jacobi U, Surber C, Weigmann HJ, Fluhr JW. The tape stripping procedure--evaluation of some critical parameters. Eur J Pharm Biopharm. 2009 Jun;72(2):317-23. doi: 10.1016/j.ejpb.2008.08.008. Epub 2008 Aug 19. PMID 18775778
- [Background] Leveque JL. EEMCO guidance for the assessment of skin topography. The European Expert Group on Efficacy Measurement of Cosmetics and other Topical Products. J Eur Acad Dermatol Venereol. 1999 Mar;12(2):103-14. PMID 10343937
- [Background] Marttin E, Neelissen-Subnel MT, De Haan FH, Bodde HE. A critical comparison of methods to quantify stratum corneum removed by tape stripping. Skin Pharmacol. 1996;9(1):69-77. doi: 10.1159/000211392. PMID 8868035
- [Background] Lemperle G, Holmes RE, Cohen SR, Lemperle SM. A classification of facial wrinkles. Plast Reconstr Surg. 2001 Nov;108(6):1735-50; discussion 1751-2. doi: 10.1097/00006534-200111000-00048. PMID 11711957
- [Background] Rieger M.M., Battista G.W. Some experiences in the safety testing of cosmetics J. Soc. Cosmet. Chem. 15:161 -172 (1964)
- [Background] Monheit GD, Gendler EC, Poff B, Fleming L, Bachtell N, Garcia E, Burkholder D. Development and validation of a 6-point grading scale in patients undergoing correction of nasolabial folds with a collagen implant. Dermatol Surg. 2010 Nov;36 Suppl 3:1809-16. doi: 10.1111/j.1524-4725.2010.01739.x. PMID 20969658
- [Background] Sachs L Applied statistics: a handbook of techniques Heidelberg: Springer, 536-539, 1981
- [Background] Salter DC, McArthur HC, Crosse JE, Dickens AD. Skin mechanics measured in vivo using torsion: a new and accurate model more sensitive to age, sex and moisturizing treatment. Int J Cosmet Sci. 1993 Oct;15(5):200-18. doi: 10.1111/j.1467-2494.1993.tb00075.x. PMID 19272125
- [Background] Serri R, Romano MC, Sparavigna A. "Quitting smoking rejuvenates the skin": results of a pilot project on smoking cessation conducted in Milan, Italy. Skinmed. 2010 Jan-Feb;8(1):23-9. PMID 20839421
- [Background] Sparavigna A., Setaro M., Galbiati G. Osservazioni sull'elasticità della pelle Cosmesi Dermatologica 22:68-78, 1988
- [Background] Sparavigna A., Setaro M., A new evaluation method of skin plastoelasticity in skin Pharmacology and toxicology. Recent advances Plenum Publishing Corporation, New York, London: 295-298, 1990
- [Background] Sparavigna A., Galbiati G. La plastoelasticità cutanea: Metodi di indagine e significato clinico Cronica Dermatologica 4: 509-517, 1992
- [Background] Sparavigna A., Setaro M. Misurazione delle proprietà meccaniche della cute mediante metodi di torsione In:"Diagnostica non invasiva in dermatologia" A cura di Stefania Seidenari, EDRA Medical Publishing & New Media, Milano, 1998, 323-328
- [Background] Sparavigna A., Setaro M. Elasticità della pelle La Pelle: Dermatologia, anno 14, mag-giu (5) 2009
- [Background] Sparavigna A, Di Pietro A, Setaro M. 'Healthy skin': significance and results of an Italian study on healthy population with particular regard to 'sensitive' skin. Int J Cosmet Sci. 2005 Dec;27(6):327-31. doi: 10.1111/j.1467-2494.2005.00287.x. PMID 18492170
- [Background] Setaro M., Sparavigna A. Is it possible to define a biological age of the skin? Preprints of 1st Joint Meeting: 14th International Congress for Bioengineering and the Skin and 8th Congress of the International Society for Skin Imaging. May 21-24, 2003, Hamburg, Germany
- [Background] Serup J, Agner T. Colorimetric quantification of erythema--a comparison of two colorimeters (Lange Micro Color and Minolta Chroma Meter CR-200) with a clinical scoring scheme and laser-Doppler flowmetry. Clin Exp Dermatol. 1990 Jul;15(4):267-72. doi: 10.1111/j.1365-2230.1990.tb02087.x. PMID 2208776
- [Background] Taelman M-C, Dederen J. C. Relative performance testing of formulations: emulsifiers Cosmetics &Toiletries magazine August 2000; 115: 37-42
- [Background] Takiwaki H. Measurement of skin color: practical application and theoretical considerations. J Med Invest. 1998 Feb;44(3-4):121-6. PMID 9597799
- [Background] Tagami H, Ohi M, Iwatsuki K, Kanamaru Y, Yamada M, Ichijo B. Evaluation of the skin surface hydration in vivo by electrical measurement. J Invest Dermatol. 1980 Dec;75(6):500-7. doi: 10.1111/1523-1747.ep12524316. No abstract available. PMID 7441001
- [Background] Weigmann H, Lademann J, Meffert H, Schaefer H, Sterry W. Determination of the horny layer profile by tape stripping in combination with optical spectroscopy in the visible range as a prerequisite to quantify percutaneous absorption. Skin Pharmacol Appl Skin Physiol. 1999 Jan-Apr;12(1-2):34-45. doi: 10.1159/000029844. PMID 10325582
- [Background] Wilhelm KP, Elsner P, Berardesca E, Maibach HI Bioengineering of the skin: Skin surface imaging and analysis CRC Press, Boca Raton, 1997
- See also: Investigation Center — http://www.derming.com
- See also: Sponsor — http://www.giulianipharma.com/